CLINICAL TRIAL: NCT07377513
Title: Follow-up Compliance for Medically Managed Corneal Ulcer Patients With SMS Reminders in a Tertiary Eye Care Setting in Western Nepal: A Quasi Experimental Study
Brief Title: Follow-up Compliance for Corneal Ulcer Patients With SMS Reminder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seva Canada Society (Other)
Collaborators: Lumbini Eye Institute and Research Centre (Other); Pragyaan Sustainable Health Outcomes Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LEIRC/ORCB/2/14122025
Record Dates: First submitted 2026-01-21; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Corneal Ulcer
Keywords: Corneal ulcer; Follow-up compliance; SMS reminder
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS reminder group (Experimental)
  Interventions: Other: SMS reminder
- Control group (No Intervention)

INTERVENTIONS:
Other: SMS reminder — Patients presenting on Monday, Wednesday, and Friday for the first time for treatment will be recruited in the intervention group.
  For those who are recruited after receiving informed consent, SMS reminders before scheduled follow-up will be sent from the hospital regarding the next scheduled visit. In addition, routine counselling will be done during the first visit regarding the follow-up schedule.
  Arms: SMS reminder group

SUMMARY:
Corneal ulcer is defined as the loss of corneal epithelium with underlying stromal infiltration and suppuration, accompanied by signs of inflammation, with or without hypopyon1. The condition may be caused by bacterial, fungal, viral or parasitic pathogens and carries a significant risk of corneal perforation and subsequent visual impairment2. These risks highlight the importance of timely treatment plans and consistent referral networks3.

A lot of patients choose to self-medicate and postpone seeking professional assistance due either their lack of awareness or forgetfulness, which results in inadequate follow-up compliance4,5. Scheduling appointments regularly is still a significant barrier to successful treatment and visual recovery.

SMS reminders have shown encouraging real-world success in improving follow-up attendance with in ophthalmology. Mobile health tools, such as the peek Community Eye Health system, have proven increased follow-up rates and improved access to eye care services in low-resource setting through automated appointment reminders and patient monitoring6.

The aim of this operational research study to evaluated the feasibility, scalability, and effectiveness of SMS reminders in improving follow-up compliance among patients with corneal ulcer at the Lumbini Eye Institute and Research Center (LEIRC), Western Nepal. The findings are expected to inform the integration of cost-effective digital health strategies to strengthen patient adherence, optimize clinical outcomes, and support eye health programs in resource limited environments.

DETAILED DESCRIPTION:
Corneal ulcer is defined as a loss of the corneal epithelium with underlying stromal infiltration and suppuration associated with the signs of inflammation with or without hypopyon1 The causative agent can be bacterial, fungal, viral, or parasitic. The causative agents of the corneal ulcer may vary depending upon the mode of injury. Fungal keratitis is endemic in tropical regions, accounting for as many as half of all corneal ulcer2 Collagenolytic and inflammatory substance, along with increased corneal matrix, metalloproteinase (MMP) activity, can lead to degradation of corneal collagen and may cause complication such as, scarring, thinning, and corneal perforation. MMPS is over-expressed in infective keratitis. Corticosteroid or tetracyclines, particular doxycycline, are used as adjuvants to antimicrobials, which help to reduce the excessive deterioration and inflammation of the corneal layers caused by corneal MMPs and reduce the inflammatory cell recruitment and infiltration3.

Corneal ulcers have a higher risk of corneal perforation. As a result, standardized referral and treatment protocols for patients with corneal ulcers are required. Potentially sight threatening corneal ulcers are at significantly higher risk for best spectacle corrected visual acuity (BSCVA) loss compared to rarely sight threatening corneal ulcers.7 Most patients use self-medication, and had delayed seeking of professional medical care4 due to a lack of awareness or simply forgetting. These factors may have contributed to the low rate of follow-up visits. Continuous education of patients and professionals is required to reduce the rate and severity of infective keratitis5. . It is a potentially vision threatening ocular emergency8 In developing countries, the average cost for accessing and receiving care for patients with corneal ulcers is US$85.8 ± 4.6 (95% confidence interval: US$76.4, 94.6). The mean total cost to diagnose and appropriately treat 1 case of keratitis such that the patient had vision better than 6/18 at final follow-up was US$56.2 ± 3.6 (95% confidence interval: US$49.0, 63.3)6 SMS reminders have demonstrated real-world success in improving follow-up adherence in ophthalmology. A study in a London ophthalmology outpatient clinic found that sending SMS reminders reduced non-attendance by 38% (relative risk of non-attendance = 0.62; 95% CI 0.48-0.80) compared to no reminder9. Additionally, broader evidence supports that SMS reminders significantly enhance follow-up adherence across healthcare contexts-meta-analysis shows pooled odds ratio (OR) for SMS improving follow-up is 1.76 (95% CI 1.37-2.26; p < 0.01) compared to controls10.In ophthalmology programs in low-resource areas, mobile health tools integrating SMS reminders have shown promising improvements. For example, the Peek Community Eye Health system, which used SMS to remind referred patients about follow-up appointments, demonstrated improved access to eye care services in rural settings11 through better attendance and tracking. Similar study protocol was designed by Bharatpur Eye Hospital to find out if counseling and reminder using SMS text messages and phone calls would boost the follow-up rates of <16 paediatric patients. 10

Given the high burden of corneal ulcers, potential for severe complications from poor follow-up, and promising evidence for SMS-based reminder systems in eye care adherence, it is necessary to study further to find the usefulness of reminder system in corneal ulcer patients. This operational research study thus aims to evaluate the feasibility, scalability, and effectiveness of SMS reminders in improving follow-up compliance among corneal ulcer patients at the Lumbini Eye Institute and Research Center, Western Nepal. The findings could catalyze the implementation of the cost-effective digital health strategies for improving outcomes in eye health across resource-limited environments.

Research objectives:

Primary objective:

• To evaluate the effectiveness of addition of SMS-based reminder system to the routine counselling versus routine counselling alone in improving follow-up compliance among corneal ulcer patients at a tertiary eye care center in western Nepal.

Secondary objectives:

• To estimate the cost-effectiveness of implementing SMS-based reminders for improving compliance.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients (18 to 70 years) of corneal ulcer in one or both eye, who are medically managed, visiting the OPD at LEIRC and have access to a mobile phone.

Exclusion Criteria:

* Less than 18 years or more than 70 years Patients who do not have a access to a mobile phone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Follow-up compliance | 6 months
  Proportion of patients who comply with scheduled follow-up visits during the study period

SECONDARY OUTCOMES:
Cost effectiveness | 6 months
  Direct and indirect cost of the SMS and routine counselling services.

IPD SHARING:
Plan to Share IPD: No